CLINICAL TRIAL: NCT02929485
Title: Dopaminergic Modulation of Frontostriatal Function With a Dopamine Agonist and COMT Inhibitor
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2011-11-3748
Record Dates: First submitted 2016-09-28; First posted 2016-10-11 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Addiction
MeSH Terms: conditions — Behavior, Addictive | interventions — Tolcapone; Bromocriptine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental: Tolcapone (Experimental): Drug: Tolcapone 200mg (single dose) administered at study visit
  Interventions: Drug: Tolcapone
- Comparator: Placebo (Placebo Comparator): Drug: Placebo for tolcapone administered at study visit
  Interventions: Drug: Placebo
- Experimental: Bromocriptine (Experimental): Drug: Bromocriptine 1.25mg (single dose) administered at study visit
  Interventions: Drug: Bromocriptine

INTERVENTIONS:
Drug: Tolcapone — Tolcapone 200mg (single dose) administered at study visit
  Other Names: Tasmar
  Arms: Experimental: Tolcapone
Drug: Placebo — Placebo (200mg) administered at study visit
  Arms: Comparator: Placebo
Drug: Bromocriptine — Drug: Bromocriptine 1.25 mg (single dose) administered at study visit
  Other Names: Parlodel
  Arms: Experimental: Bromocriptine

SUMMARY:
In this study, the investigators are looking at how people make decisions about reward-related items, both monetary and food related after taking either the dopamine agonist bromocriptine or the COMT inhibitor tolcapone, in healthy control subjects. Subjects will fill self-report questionnaires and undergo an MRI scan.

DETAILED DESCRIPTION:
The investigators aim to understand how the brain's dopamine system impacts monetary and food-related decision making. The investigators aim to use tolcapone and bromocriptine due to the temporary change in the levels of dopamine in the brain. The investigators also aim to determine if genetics, personality traits, or a family history of alcoholism change how these drugs affect decision making.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years.
* Subject is right-handed.
* If female, subject is non-lactating, not pregnant, and using a reliable contraception method (i.e. abstinence, intrauterine device (IUD), hormonal birth control or barrier method).
* Subject is able to read and speak English.
* Subject is a high school graduate.
* Subject is able and willing to provide written and informed consent.
* Subject is able to understand and follow the instructions of the investigator, and understand all ratings scales.
* Subject is in good health.

Exclusion Criteria

* Using cocaine, stimulants (other than THC, nicotine, & caffeine)amphetamines, hallucinogens, "ecstasy", opiates, sedatives, pain pills, sleeping pills or other psychoactive drugs within two weeks of the start of the study OR more than 10 times in the last year.
* Has a current dependence on, or addiction to any psychoactive drug (except nicotine or caffeine) including alcohol.
* Clinically significant medical or psychiatric illness requiring treatment as determined by screening blood tests, medical history, and physical exam performed or reviewed by the study physician.
* Subject has a history of major alcohol related complications within the proceeding 2 years (liver failure/cirrhosis, pancreatitis, esophageal varices, etc.)
* Liver function test ≥ 3 times normal upper limit.
* BAC level > 0.05% at the beginning of screening visit (within margin of error of detection).
* Has a neurological dysfunction or psychiatric disorder.
* Has severe low blood pressure.
* Has uncontrolled high blood pressure.
* Regular use of any of the drugs on the tolcapone or entacapone contraindications list OR within 2 weeks of drug administration.
* Regular use of SSRIs.
* Has an allergy or intolerance to tolcapone or entacapone.
* Subject has received an investigational drug within 30 days of screening visit.
* Subject is considered unsuitable for the study in the opinion of the investigator or study physician for any other reason.

MRI Exclusion Criteria:

* The subject has metal (metal plates, pins, wires or screws, artificial limb, joint replacement or anything that might have been inserted during an operation) in his/her body.
* Subject has a pacemaker, defibrillator, stent, or any metal implants related to heart/blood flow problems.
* Subject has worked with metals (ie. metallurgy, metal shaving, welding, soldering, etc).
* Subject has been wounded with anything metal (bullet, shrapnel or metal filling).
* Has ever gotten a piece of metal in the eye.
* Has tattoos done with ink containing metal or permanent eyeliner.
* Wears color contact lenses.
* Has a hearing problem or hearing aid, cochlear implant or past ear surgery.
* Has any irremovable dental bridges, dental plates, metal caps or any other non-removable metal in the mouth.
* The subject is claustrophobic.
* The subject is pregnant. (women only)
* Has a IUD. (women only)
* Significantly overweight.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07 (Estimated); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-01-31 (Estimated)

PRIMARY OUTCOMES:
Measure Effects of Placebo,Tolcapone, Bromocriptine on Reaction Time | 3 weeks
  Participants will play the Dictator Game. Behavioral responses to the game during each arm (placebo, tolcapone, and bromocriptine) will be measured by subject reaction time .
Measure Effects of Placebo,Tolcapone, Bromocriptine on Accuracy | 3 weeks
  Participants will play the Dictator Game. Behavioral responses to the game during each arm (placebo, tolcapone, and bromocriptine) will be measured by subject accuracy (correct or incorrect responses).

SECONDARY OUTCOMES:
Measure Observed Changes in Resting State Neural Activity | 3 weeks
  Resting-state data will be processed off-line using neuroimaging analysis software according to standard procedures for image slice-timing correction, realignment, normalization and smoothing. Changes in regional brain activity will be measured during the placebo, tolcapone and bromocriptine conditions.
Measure Observed Changes in Task Dependent Neural Activity | 3 weeks
  Task dependent fMRI data will be processed off-line using neuroimaging analysis software according to standard procedures for image slice-timing correction, realignment, normalization and smoothing. Changes in task dependent brain activity will be measured during the placebo, tolcapone and bromocriptine conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kayser, MD,PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, Berkeley, Berkeley, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No